CLINICAL TRIAL: NCT05875285
Title: Methotrexate Iontophoresis Versus Coal Tar Ointement in the Treatment of Primary Palmer Hyper Hidrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nayera Radwan Fathy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nayera_Radwan_2023
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Hyperhidrosis; Iontophore
MeSH Terms: conditions — Hyperhidrosis | interventions — Iontophoresis; Methotrexate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotreaxate iontophoresis (Experimental): Thirty patients of both sexes of primary palmar hyperhidrosis are selected to participate in this group from EL KASR EL- AINI
  Interventions: Other: Iontophoresis with methotrexate
- Coal tar ointment (Experimental): Thirty patients of both sexes of primary palmar hyperhidrosis are selected to participate in this group from EL KASR EL- AINI
  Interventions: Other: Iontophoresis with coal tar ointement

INTERVENTIONS:
Other: Iontophoresis with methotrexate — The methotrexate iontophoresis group the patient's hands are placed in direct contact with the conductive electrodes.
  The patient will receive full explanation to the purpose of the treatment, the therapeutic and physiological benefits of this method of treatment. Before starting the treatment, all the previous measurements of each patient in this group is taken for a comparison.
  Every patient will receive 12 sessions 3times/week every session consist of 30 minutes application of methotrexate iontophoresis using continuous direct current, the patient should feel mild tingling sensation (not painful), the polarity should be reversed halftime of treatment session, as the anodal current is more effective.
  Arms: Methotreaxate iontophoresis
Other: Iontophoresis with coal tar ointement — For coal tar ointement group the ointement is putted direct on the skin after describing the instruction and method of application and time of application and do alarm instead not to forget.
  Arms: Coal tar ointment

SUMMARY:
The purpose of the study is to compare the therapeutic effect of methotrexate iontophoresis versus coal tar ointment on the the treatment of primary palmer hyperhidrosis?

DETAILED DESCRIPTION:
Some researchers stated that hyperhidrosis can render the skin susceptible to infection because of the continuous dampness of the skin. The condition may become socially, psychologically and professionally debilitating.

There are a lot of literatures concerned with studying the modalities used in the treatment of primary palmar hyperhidrosis, so this study will be conducted to compare between two of them and to show the best one for treating primary palmar hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary palmar hyperhidrosis to extend that their palms are wet during most of the day (score 3 and 4 in the Hyperhidrosis Disease Severity Scale) was included in this study.
* The palmer hyperhidrosis patient's age ranged from 15 to 35 years.
* All patients will be examined by dermatologist before starting the study.

Exclusion Criteria:

The study excluded the following patients:

* Patients with medical conditions that associated with hyperhidrosis are excluded, these conditions include:- hyperthyroidism, diabetes mellitus, parkinsonism, spinal cord injury, brain damage, congestive heart failure, anxiety, alcoholism and menopause.
* Patients who received any treatment with a drug that was affecting sweating e.g. (thyroxin, anxiolytics…..) that is not stopped at least 4 weeks preceding the study.
* Patients with cardiac conditions such as arrhythmia, ischemic heart disease, low exercise tolerance, low respiratory reserve were excluded.
* Patients, who have a local wound, sever eczema and severe fungal infection of the palms to minimize risk of local burn.
* Patients who have sensory disorders.
* Female patients who are pregnant and lactating.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-08-20 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in Sweat output | at baseline and after 4 weeks of intervention
  Sweat output was objectively measured by recording mass gained by a standard diaper of approximately 30gm that was placed in contact with palms for 10 minutes and then was weighted using laboratory mass scale
Assessing the change in degree of severity of hyperhidrosis | at baseline and after 4 weeks of intervention
  By using Hyperhidrosis disease severity scale. It is a (4) points scale that is used to determine the degree of severity of hyperhidrosis

CONTACTS AND LOCATIONS:
Overall Officials: Nayera Radwan, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physical therapy cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No